CLINICAL TRIAL: NCT02646631
Title: Behavioral and Educational Tools to Improve Epilepsy Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-01386
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Usual Treatment (Experimental)
  Interventions: Other: Usual Care; Other: Educational Materials
- MORE (Experimental)
  Interventions: Other: Usual Care; Behavioral: Management of Risks in Epilepsy (MORE); Other: Educational Materials
- MORE + MI (Active Comparator)
  Interventions: Other: Usual Care; Behavioral: Management of Risks in Epilepsy (MORE); Behavioral: Telephone-based motivational interviewing (MORE+MI); Other: Educational Materials

INTERVENTIONS:
Other: Usual Care — Participants assigned to this treatment will receive the usual care as determined by their physician
Behavioral: Management of Risks in Epilepsy (MORE) — MORE is a smartphone application which participants use to record information on a daily basis about seizures (severity, type), medications, and mood and stress levels. It also includes a camera-based application which uses a pill scanner and photo to record the identity and quantity (dose) of medications just prior to them being taken. Also included in the app are medication reminders, educational video clips, and self-management tips.
  Arms: MORE; MORE + MI
Behavioral: Telephone-based motivational interviewing (MORE+MI) — Participants will receive a total of 4 motivational interviewing sessions over the phone. These sessions last approximately 20 minutes each and build on the educational materials already provided within the MORE app.
  Arms: MORE + MI
Other: Educational Materials — Printed educational materials on the management of epilepsy

SUMMARY:
The long-term goal of this research is to improve seizure control among patients with epilepsy, which has the potential to improve quality of life for thousands of people living with epilepsy and reduce health care utilization, social and economic costs, and epilepsy-related mortalities. Participants who are suffering from epilepsy will be randomized to receive usual care (UC), a smartphone-based self-management intervention called Management of Risks in Epilepsy (MORE), or MORE + telephone-based motivational interviewing (MI). Participants will be followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. English- or Spanish-speaking
3. Partial (focal) or generalized epilepsy (as confirmed with epileptiform activity on an electroencephalogram)
4. Poor medication adherence
5. Willing and able to use a smartphone (provided by the study) to manage disease.

Exclusion Criteria:

1. Known or suspected psychogenic nonepileptic seizures as sole seizure type
2. Active psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Percent adherence to anti-epileptic drug schedule (pill counts) | 3 months

SECONDARY OUTCOMES:
Number of patients who complete the study | 3 months
Percentage of MI sessions completed | 3 months
Percentage of diary entries completed | 3 months
Adherence to anti-epileptic drug schedule (self-reported) as measured by the Morisky Medication Adherence Scale | 3 months
  As measured by the Morisky Medication Adherence Scale
Seizure frequency | 3 months
Quality of life as measured by the Quality of Life in Epilepsy questionnaire score | 3 months
Quality of life as measured by the PROMIS-10 questionnaire score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Spruill, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States